CLINICAL TRIAL: NCT02102425
Title: Effects by Omission of Bandage Over Exit Site at Patients in Peritoneal Dialysis (PD).Randomized Controlled Cross-over Study
Brief Title: Effects by Omission of Bandage Over Exit Site
Acronym: EXIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Edith Mark (Other)
Collaborators: Aalborg University Hospital (Other)
Responsible Party: Sponsor-Investigator, Edith Mark, Postdoc in Clinical Nursing, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Other Study IDs: N-20130076
Record Dates: First submitted 2014-03-20; First posted 2014-04-03 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Renal Insufficiency, Chronic
Keywords: Peritoneal Dialysis; Exit site infection; Exit site care; Bandage; Prevention; Guidelines
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Chronic kidney disease, PD: Patients with or without bandage over exit site
  Interventions: Procedure: Patients with or without bandage over exit site

INTERVENTIONS:
Procedure: Patients with or without bandage over exit site

SUMMARY:
Peritoneal dialysis, known as p- dialysis (PD), is a dialysis form in which the blood is purified by using the body's peritoneum. PD dependents on good access to peritoneum. For this, a catheter is implanted in the peritoneum and tunneled 2-3 cm below the skin. The way out is called exit site and is close to the navel.

Patients are selected at random to use bandage or not use bandage for three months, then cross-over. The overall objective of the research is that the patient in PD maintains a complete and healthy skin without signs of infection around the exit site. In the study effects by omission of bandage over exit site at patients in PD are examined when the patients are in a stable process with PD. The patient's exit site is assessed according to skin character and examined for infection.

The hypothesis is that there is no greater rate of infection in patients without bandage than in patients with bandage over the exit site, and that patients without bandage will have stronger skin around exit site.

DETAILED DESCRIPTION:
Background: For a patient in a stable (PD) there is no evidence for using bandage over exit site. Guidelines refer to this as an unsolved question.

An exit site infection can lead to tunnel infection and to peritonitis, which can be fatal. For this reason it is very important to prevent exit site infections and at the same time it is very important to reduce antibiotic which is a general problem in health care. (In Denmark, the patient does not use antibiotic cream around exit site, preventive.) Few years back, the care of the exit site was associated with sterile techniques, and the use of bandage was an obligatory procedure. The risk of infection appears now to be much less than first thought, but it is unclear what procedures are best: bandage or no bandage.

At present, most patients use bandage, but some patients drop it when bandage leads to maceration of the skin, allergy or wetness around the exit site. Other patients simply do not want to use bandage with subjective reasons. A dialysis catheter interferes with the patient's bodily life, integrity, autonomy and with the social sphere.

The nurses in the PD clinic at Aalborg University Hospital might have observed that patients without bandage do not get more infections around the exit site in relation to the patients using bandage. However, the study should develop evidence guidelines.

Objective: The aim of the study is to study the effects by omission of bandage over exit site at patient in PD when the patient is in a stable course. The purpose is that the patient maintains an unbroken skin without signs of infection around the exit site.

Design: Randomized controlled cross-over study. Setting: Department of outpatient clinic for peritoneal dialysis, Departments of Nephrology, Aalborg University Hospital in Region Northern Denmark.

Participants: The estimated numbers of participants are 35 men and women aged > 18 years. The patients are in stable PD with uraemia chronic classified by International Statistical Classification of Diseases and Related Health Problems, Tenth Revision (ICD10) - kode DN189 - and will be enrolling and included by invitations in the outpatient clinic. Exclusion criteria: special reasons for protection of the exit site - eg. critical illness, stay in areas with high risk of infection or body movements that require special fixation of the exit site, do not understand or speak Danish, mental impairment or symptoms of eczema around the exit site.

Inclusion time: March 2014 to september 2015. Method: By inclusion patients are randomized to either use or not use bandage. After 3 months the patient will cross over and do the opposite.

By inclusion investigators collect data to baseline characteristics (age, sex, marital status, other diseases, smoking, height and weight, medication use, self-reliance, time of construction of p-catheter, type of catheter, who is caring for the exit site at home and how often is changing of bandage per. week, previous infections, skin itching). The nurse in the outpatient clinic also examines a bath instruction with the patient.

The primary endpoint is the condition of the skin around the exit site as measured by Sunnybrook PD Catheter Exit Site Assessment Tool prepared by Patsy Cho and colleagues. Following parameters are recorded: Redness, crust, swelling, pain, secretion. The patient is assessed a total of five times with this skin assessment: at inclusion, after 6 weeks, 3 months (cross-over), 4.5 months and 6 months.

At these four controls investigators also collect data on: Infection, self-reliance, who is caring for the exit site and how often is changing of bandage per. week, skin itching. Moreover, the patient must answer a questionnaire on compliance and experiences of wearing bandage or not wearing bandage.

All data entered in a database. Main outcome measures: The primary endpoint is the condition of the skin around the exit site. The secondary endpoints will partly be the number of exit site infections, tunnel infections and peritonitis and the third point is a record of patient compliance and experiences in relation to participation in the project.

The trial is approved by the local Ethics Committee, registration number: N-20130076

ELIGIBILITY:
Inclusion Criteria:

Patients with uraemia chronic classified by ICD10 kode DN189. The patients are in stable PD. Talk og understand Danish.

Exclusion Criteria:

Special reasons for protection of the exit site (- eg. critical illness, stay in areas with high risk of infection or body movements that require special fixation of the exit site) Mental impairment.

Symptoms of eczema around the exit site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nurses in the PD clinic at Aalborg University Hospital might have observed that patients without bandage do not get more infections around the exit site in relation to the patients using bandage. However, the study should develop evidence guidelines.
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-10 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Healthy unbroken skin | The patient is assessed after 6 months.
  The primary endpoint is the condition of the skin around the exit site as measured by Sunnybrook PD Catheter Exit Site Assessment Tool prepared by Patsy Cho and colleagues. Following parameters are recorded: Redness, crust, swelling, pain, secretion.

SECONDARY OUTCOMES:
Infection | The patient is assessed efter 6 months
  Signs of infection are continuously monitored both by the patient and the nursing staff at the controls. Patients can always contact the staff on suspicion of infection. By an infection the patient is deleted temporarily the study. Once the infection is successfully completed, the patient can enter the the study again

OTHER OUTCOMES:
Patient's experience of the exit site with or without bandage | Questionnaire after 6 months
  The patient's subjective feelings and experience of the exit site and bandage examined through a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Erik E Sørensen, PhD Nursing, Study Chair — Clinical Nursing Research Unit, Aalborg University Hospital, Denmark
Locations (1):
- PD-ambulatorium, Clinical Nursing Research Unit/Department of Nephrology, Aalborg University Hospital,, Aalborg, Denmark

REFERENCES:
- See also: Clinical Nursing Research Unit, Aalborg University Hospital, Denmark — http://www.foksy.dk